CLINICAL TRIAL: NCT03956940
Title: A Sorafenib-Regorafenib Sequence Treatment Monitoring Study Using Liquid Biopsy
Brief Title: Analysis of cfDNA in Patients With Hepatocarcinoma and Treated by Sorafenib or Regorafenib
Acronym: HELP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of the scientific and medical context that is no longer favorable to our study. This has resulted in the termination of inclusions.
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A02911-54
Record Dates: First submitted 2019-05-15; First posted 2019-05-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Hepatocarcinoma
Keywords: Hepatocarcinoma; cfDNA; intplex
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intplex test (Experimental): In vitro diagnostic device
  Interventions: Device: Intplex test

INTERVENTIONS:
Device: Intplex test — Blood sample at baseline, 15 days, 4-8-16 weeks and then every 12 weeks

SUMMARY:
The aim of this trial is to investigate whether quantitative analysis of the total concentration of circulating free deoxyribonucleic acid (cfDNA) and of the cfDNA integrity index (DII) (Intplex®) may reflect hepatocellular carcinoma (HCC) tumor dynamics or response for patients treated by Sorafenib or Regorafenib and if it could be used as a tool for patient management under targeted therapy.

DETAILED DESCRIPTION:
Circulating free deoxyribonucleic acid (cfDNA) is increasingly used in oncology with the aiml of early diagnosis of the disease, its therapeutic management and monitoring the evolution of the disease. Numerous publications have shown that the cfDNA concentration is correlated with the pathology of cancer. Larger amounts of cfDNA are detected in metastatic patients or patients with advanced cancer. However, the cfDNA concentrations have not yet shown their clinical interest mainly because of the variations in the same individual during the effort or the moment of collection of the blood sample. The concept of the integrity of cfDNA has also been studied as a biomarker in oncology and seems to show an interesting clinical value. The cfDNA is essentially released by cell apoptosis generating 170 bp fragments, corresponding to the size of a nucleosome. Many studies have shown that the integrity of cfDNA increases with the pathology of cancer. Thus, tumor-derived cfDNA is more fragmented than healthy cells with fragments smaller than the size nucleosome.

To date, no predictive biomarker is available for the management of treatment with Sorafenib which is a targeted therapy with a marketing authorization in first-line treatment of HCC (hepatocellular carcinoma) or second line with Regorafenib, treatment having shown a benefit positive on overall survival in the Resorce study. AFP (alpha-foetoprotein) is the only serum marker available with an inconstant increase in patients with HCC in fact only 30 to 40% of patients have abnormal values. In liver cancer, Ono et al showed that serum cfDNA is positively correlated with a larger tumor size.

This study shows that the rate of tumor cfDNA reflects the progression of the disease. Jiang et al showed that cfDNA derived from HCC is more fragmented than that derived from healthy cells, with fragments smaller than the size nucleosome.

These data demonstrate the potential utility of cfDNA amount and integrity as a biomarker for individualized management of hepatocellular carcinoma.

This new marker is expected to be an effective tool to overcome the lack of specificity of the AFP (alpha foetoprotein) assay in this pathology.

The investigator's team developed an Intplex® test that showed significant discrimination between healthy individuals and cancer patients.

The aim of this trial is to investigate whether quantitative analysis of the total concentration of cfDNA and of the cfDNA integrity index (DII) (Intplex®) may reflect HCC tumor dynamics or response for patients treated by Sorafenib or Regorafenib and if it could be used as a tool for patient management under targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Histological or cytological documentation of hepatocellular carcinoma (HCC) or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases (AASLD) criteria in patients with a confirmed diagnosis of cirrhosis
3. Patient treated for stage B hepatocellular carcinoma (multifocal disease) or stage C (metastatic disease) according to Barcelona Clinic liver cancer, regardless of treatment line, and that cannot benefit from local treatments such as resection, local ablation, chemoembolization
4. At least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST criteria 1.1 and modified RECIST for HCC
5. Liver function status Child-Pugh Class A
6. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory tests:

   * Hemoglobin > 8.5 g/dL
   * Absolute neutrophil count ≥ 1500/mm3
   * Platelet count ≥ 60,000/ mm3
   * Total bilirubin ≤ 2 mg/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN)
   * Serum creatinine ≤ 1.5 x Upper limit normal (ULN)
   * Lipase ≤ 2 x ULN
   * Prothrombin time-international normalized ratio (PT-INR) < 2.3 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN
   * Glomerular Filtration Rate (GFR) ≥ 30 mL/min/1.73 m2
8. Life expectancy ≥ 3 months
9. Women of childbearing potential and men must agree to use adequate contraception
10. Patients must be affiliated to a Social Security System
11. Written informed consent signed

    Patients initially treated with Sorafenib, will be switched to Regorafenib if all the above conditions are still met and, in addition:
12. Documented progression under treatment with Sorafenib (defined as documented radiological and/or clinical and/or biological progression)

Exclusion Criteria:

1. Prior liver transplantation or candidates for liver transplantation
2. Hypersensitivity to the active substance or to any of the excipients
3. Patients with large esophageal varices at risk of bleeding that are not being treated with conventional medical intervention
4. Past or concurrent history of neoplasm other than HCC, except for in situ carcinoma of the cervix uteri and/or non-melanoma skin cancer and superficial bladder tumors. Any cancer curatively treated > 3 years prior to study entry is permitted
5. Known history or symptomatic metastatic brain or meningeal tumors
6. Major surgical procedure or significant traumatic injury within 28 days before enrollment
7. Congestive heart failure New York Heart Association (NYHA) ≥ class 2
8. Unstable angina or myocardial infarction within the past 6 months before enrollment
9. Cardiac arrhythmias requiring anti-arrhythmic therapy
10. Uncontrolled hypertension
11. Patients with phaeochromocytoma
12. Uncontrolled ascites
13. Persistent proteinuria of NCI-CTCAE version 4.0 ≥ Grade 3
14. Ongoing infection > Grade 2 according to NCI-CTCAE version 4.0. Hepatitis B is allowed if no active replication is required
15. Clinically significant bleeding NCI-CTCAE version 4.0 ≥ Grade 3 within 30 days before enrollment
16. Arterial or venous thrombotic or embolic events such as cerebrovascular accident, deep vein thrombosis or pulmonary embolism within 6 months before enrollment
17. Any psychological, familial, sociological, geographical or illness or medical condition that could jeopardize the safety of the patient and/or his compliance with the study protocol and follow-up procedure
18. Known history of human immunodeficiency virus (HIV) infection
19. Seizure disorder requiring medication
20. Non-healing wound, ulcer or bone fracture
21. Active autoimmune disease (lupus, sclerodermia, rheumatoid arthritis, …)
22. Any malabsorption condition
23. Breast feeding
24. Pregnancy
25. High performance sport practice
26. Patient unable to swallow oral medication

    Patients who discontinue sorafenib will not be switched to regorafenib if any of the condition listed above occurs and/or the following criteria are met:
27. Prior discontinuation of prior Sorafenib therapy due to Sorafenib-related toxicity
28. Unresolved toxicity (Sorafenib) ≥ NCI-CTCAE version 4.0 Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of total circulating free deoxyribonucleic acid (cfDNA) concentration at the baseline. | Baseline
  Total cfDNA concentration is considered as detected if total cfDNA concentration ≥ 5 ng/mL and not detected if total cfDNA concentration < 5 ng/mL

SECONDARY OUTCOMES:
total circulating free deoxyribonucleic acid (cfDNA) fragmentation index | Baseline
  Fragmentation of cfDNA
Objective response rate | Approximately 36 months
  From the date of inclusion to the date of death from any cause
Disease control rate | Approximately 36 months
  From the date of inclusion to the date of death from any cause
Progression-Free Survival | Approximately 36 months
  The time from the date of start of Sorafenib (Regorafenib respectively) to the date of first documented
Time-to-progression | Approximately 36 months
  The time from the date of start of Sorafenib (Regorafenib respectively) to the date of first documented progression ( radiological or clinical)
Overall Survival | Approximately 36 months
  The time from the date of start of Sorafenib to the date of documented death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Eric ASSENAT, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (6):
- France (6):
  - Hôpital Saint-Eloi, Montpellier, Hérault
  - CHU Grenoble - Hôpital Michalon, Grenoble, Isère
  - Hôpital Hôtel Dieu, Nantes, Loire-Atlantique
  - CHRU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHRU de Lille - Hôpital Claude Duriez, Lille, Nord
  - Hôpital Beaujon, Clichy, Seine-Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta S, Bent S, Kohlwes J. Test characteristics of alpha-fetoprotein for detecting hepatocellular carcinoma in patients with hepatitis C. A systematic review and critical analysis. Ann Intern Med. 2003 Jul 1;139(1):46-50. doi: 10.7326/0003-4819-139-1-200307010-00012. PMID 12834318
- [Background] Riaz A, Ryu RK, Kulik LM, Mulcahy MF, Lewandowski RJ, Minocha J, Ibrahim SM, Sato KT, Baker T, Miller FH, Newman S, Omary R, Abecassis M, Benson AB 3rd, Salem R. Alpha-fetoprotein response after locoregional therapy for hepatocellular carcinoma: oncologic marker of radiologic response, progression, and survival. J Clin Oncol. 2009 Dec 1;27(34):5734-42. doi: 10.1200/JCO.2009.23.1282. Epub 2009 Oct 5. PMID 19805671
- [Background] Chan SL, Mo FK, Johnson PJ, Hui EP, Ma BB, Ho WM, Lam KC, Chan AT, Mok TS, Yeo W. New utility of an old marker: serial alpha-fetoprotein measurement in predicting radiologic response and survival of patients with hepatocellular carcinoma undergoing systemic chemotherapy. J Clin Oncol. 2009 Jan 20;27(3):446-52. doi: 10.1200/JCO.2008.18.8151. Epub 2008 Dec 8. PMID 19064965
- [Background] Duvoux C, Roudot-Thoraval F, Decaens T, Pessione F, Badran H, Piardi T, Francoz C, Compagnon P, Vanlemmens C, Dumortier J, Dharancy S, Gugenheim J, Bernard PH, Adam R, Radenne S, Muscari F, Conti F, Hardwigsen J, Pageaux GP, Chazouilleres O, Salame E, Hilleret MN, Lebray P, Abergel A, Debette-Gratien M, Kluger MD, Mallat A, Azoulay D, Cherqui D; Liver Transplantation French Study Group. Liver transplantation for hepatocellular carcinoma: a model including alpha-fetoprotein improves the performance of Milan criteria. Gastroenterology. 2012 Oct;143(4):986-94.e3; quiz e14-5. doi: 10.1053/j.gastro.2012.05.052. Epub 2012 Jun 29. PMID 22750200
- [Background] Personeni N, Bozzarelli S, Pressiani T, Rimassa L, Tronconi MC, Sclafani F, Carnaghi C, Pedicini V, Giordano L, Santoro A. Usefulness of alpha-fetoprotein response in patients treated with sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2012 Jul;57(1):101-7. doi: 10.1016/j.jhep.2012.02.016. Epub 2012 Mar 10. PMID 22414760
- [Background] Yamashita T, Forgues M, Wang W, Kim JW, Ye Q, Jia H, Budhu A, Zanetti KA, Chen Y, Qin LX, Tang ZY, Wang XW. EpCAM and alpha-fetoprotein expression defines novel prognostic subtypes of hepatocellular carcinoma. Cancer Res. 2008 Mar 1;68(5):1451-61. doi: 10.1158/0008-5472.CAN-07-6013. PMID 18316609
- [Background] Sozzi G, Conte D, Mariani L, Lo Vullo S, Roz L, Lombardo C, Pierotti MA, Tavecchio L. Analysis of circulating tumor DNA in plasma at diagnosis and during follow-up of lung cancer patients. Cancer Res. 2001 Jun 15;61(12):4675-8. PMID 11406535
- [Background] Thierry AR, Mouliere F, El Messaoudi S, Mollevi C, Lopez-Crapez E, Rolet F, Gillet B, Gongora C, Dechelotte P, Robert B, Del Rio M, Lamy PJ, Bibeau F, Nouaille M, Loriot V, Jarrousse AS, Molina F, Mathonnet M, Pezet D, Ychou M. Clinical validation of the detection of KRAS and BRAF mutations from circulating tumor DNA. Nat Med. 2014 Apr;20(4):430-5. doi: 10.1038/nm.3511. Epub 2014 Mar 23. PMID 24658074
- [Background] Thierry AR, El Messaoudi S, Gahan PB, Anker P, Stroun M. Origins, structures, and functions of circulating DNA in oncology. Cancer Metastasis Rev. 2016 Sep;35(3):347-76. doi: 10.1007/s10555-016-9629-x. PMID 27392603
- [Background] Ono A, Fujimoto A, Yamamoto Y, Akamatsu S, Hiraga N, Imamura M, Kawaoka T, Tsuge M, Abe H, Hayes CN, Miki D, Furuta M, Tsunoda T, Miyano S, Kubo M, Aikata H, Ochi H, Kawakami YI, Arihiro K, Ohdan H, Nakagawa H, Chayama K. Circulating Tumor DNA Analysis for Liver Cancers and Its Usefulness as a Liquid Biopsy. Cell Mol Gastroenterol Hepatol. 2015 Jun 17;1(5):516-534. doi: 10.1016/j.jcmgh.2015.06.009. eCollection 2015 Sep. PMID 28210698
- [Background] Jiang P, Chan CW, Chan KC, Cheng SH, Wong J, Wong VW, Wong GL, Chan SL, Mok TS, Chan HL, Lai PB, Chiu RW, Lo YM. Lengthening and shortening of plasma DNA in hepatocellular carcinoma patients. Proc Natl Acad Sci U S A. 2015 Mar 17;112(11):E1317-25. doi: 10.1073/pnas.1500076112. Epub 2015 Feb 2. PMID 25646427
- [Background] Diaz LA Jr, Bardelli A. Liquid biopsies: genotyping circulating tumor DNA. J Clin Oncol. 2014 Feb 20;32(6):579-86. doi: 10.1200/JCO.2012.45.2011. Epub 2014 Jan 21. PMID 24449238
- [Background] El Messaoudi S, Mouliere F, Du Manoir S, Bascoul-Mollevi C, Gillet B, Nouaille M, Fiess C, Crapez E, Bibeau F, Theillet C, Mazard T, Pezet D, Mathonnet M, Ychou M, Thierry AR. Circulating DNA as a Strong Multimarker Prognostic Tool for Metastatic Colorectal Cancer Patient Management Care. Clin Cancer Res. 2016 Jun 15;22(12):3067-77. doi: 10.1158/1078-0432.CCR-15-0297. Epub 2016 Feb 4. PMID 26847055
- [Background] Mouliere F, El Messaoudi S, Pang D, Dritschilo A, Thierry AR. Multi-marker analysis of circulating cell-free DNA toward personalized medicine for colorectal cancer. Mol Oncol. 2014 Jul;8(5):927-41. doi: 10.1016/j.molonc.2014.02.005. Epub 2014 Mar 24. PMID 24698732
- [Background] Zonta E, Nizard P, Taly V. Assessment of DNA Integrity, Applications for Cancer Research. Adv Clin Chem. 2015;70:197-246. doi: 10.1016/bs.acc.2015.03.002. Epub 2015 Apr 11. PMID 26231488